CLINICAL TRIAL: NCT00039078
Title: The Use of TheraSphere® for the Treatment of Unresectable Hepatocellular Carcinoma
Brief Title: Radiolabeled Glass Beads (TheraSphere®) in Treating Patients With Primary Liver Cancer That Cannot Be Removed by Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Record created in error - not a research study
Sponsor: Allan Tsung (Other)
Responsible Party: Sponsor-Investigator, Allan Tsung, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Purpose: Treatment
Other Study IDs: PCI-IRB-0611014; CDR0000069336 (Registry Identifier: PDQ (Physician Data Query)); PCI-IRB-000656; PCI-IRB-000871; NCI-V02-1701
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Liver Cancer
Keywords: localized unresectable adult primary liver cancer; recurrent adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Radiation: yttrium Y 90 glass microspheres

SUMMARY:
RATIONALE: Internal radiation therapy uses radioactive material placed directly into or near a tumor to kill tumor cells. Using radiolabeled glass beads to kill tumor cells may be effective treatment for liver cancer that cannot be removed by surgery.

PURPOSE: This phase II trial is studying the side effects of hepatic arterial infusion using yttrium-90 microspheres (TheraSphere®) to see how well it works in treating patients with liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Provide supervised access to yttrium-90 glass microspheres (TheraSphere®) for patients with unresectable hepatocellular carcinoma.
* Determine the response in patients with unresectable hepatocellular carcinoma treated with hepatic arterial infusion of yttrium-90 glass microspheres.
* Determine the toxic effects and adverse experiences associated with this therapy in these patients.
* Determine the survival time of patients treated with this therapy.
* Determine the time to progression of disease in the liver, duration of response, and progression-free interval of patients treated with this therapy.
* Evaluate the influence of pretreatment characteristics on efficacy parameters in patients treated with this therapy.
* Assess the quality of life of patients treated with this therapy.

OUTLINE: Radioactive material yttrium-90 glass microspheres (TheraSphere®) is infused directly into a liver tumor in order to kill tumor cells and cause less damage to the normal tissue. Patients receive TheraSphere® via hepatic arterial infusion on day 1. This artery is accessed through the femoral artery in the groin. This procedure is generally completed on an outpatient basis. Patients may receive a single dose to the whole liver, or sequential treatments to each side of the liver approximately 30 to 90 days apart. Patients may be re-treated at a later time.

Patients are followed every 2 to 4 months for the rest of their lives to access tumor progression, symptom management and quality of life.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of hepatocellular carcinoma (HCC)

  * Histopathology confirmation may be waived in patients with a radiographically identifiable liver mass in addition to known laboratory or clinical risk factors for HCC, and/or an elevated alpha-fetoprotein (AFP) level
* No significant extrahepatic disease that may represent an imminent life-threatening outcome
* No evidence of potential delivery of greater than 16.5 mCi (30 Gy absorbed dose) of radiotherapy to the lungs on either the first yttrium-90 glass microspheres (TheraSphere®) administration or with cumulative delivery of radiation to the lungs over multiple treatments due to any angiographically uncorrectable flow to the gastrointestinal tract

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* No hepatic dysfunction
* Bilirubin ≤ 2.0 mg/dL
* No vascular abnormalities or severe peripheral vascular disease that would preclude angiography or selective visceral catheterization
* No pulmonary insufficiency
* No evidence of detectable technetium Tc 99m macroaggregates of albumin flow to the stomach or duodenum after application of established angiographic techniques to stop such flow
* No contraindications to angiography
* No contraindications to selective visceral catheterization
* No other condition or cormorbidity that would preclude study treatment
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 30 days after study

PRIOR CONCURRENT THERAPY:

* At least 1 month since prior chemotherapy, radiotherapy, or surgery
* No other concurrent investigational agents or anticancer therapy for HCC

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2000-08; Primary Completion 2000-08; Study Completion 2000-08

PRIMARY OUTCOMES:
Response to treatment
Survival time from treatment
Adverse experiences

CONTACTS AND LOCATIONS:
Overall Officials: T. Clark Gamblin, MD, Study Chair — UPMC Cancer Center at UPMC Presbyterian
Locations (1):
- UPMC Liver Cancer Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Goin JE, Salem R, Carr BI, Dancey JE, Soulen MC, Geschwind JF, Goin K, Van Buskirk M, Thurston K. Treatment of unresectable hepatocellular carcinoma with intrahepatic yttrium 90 microspheres: a risk-stratification analysis. J Vasc Interv Radiol. 2005 Feb;16(2 Pt 1):195-203. doi: 10.1097/01.RVI.0000142602.79459.90. PMID 15713920
- [Background] Geschwind JF, Salem R, Carr BI, Soulen MC, Thurston KG, Goin KA, Van Buskirk M, Roberts CA, Goin JE. Yttrium-90 microspheres for the treatment of hepatocellular carcinoma. Gastroenterology. 2004 Nov;127(5 Suppl 1):S194-205. doi: 10.1053/j.gastro.2004.09.034. PMID 15508085
- [Background] Salem R, Thurston KG, Carr BI, Goin JE, Geschwind JF. Yttrium-90 microspheres: radiation therapy for unresectable liver cancer. J Vasc Interv Radiol. 2002 Sep;13(9 Pt 2):S223-9. doi: 10.1016/s1051-0443(07)61790-4. PMID 12354840
- [Result] Carr BI. Hepatic arterial 90Yttrium glass microspheres (Therasphere) for unresectable hepatocellular carcinoma: interim safety and survival data on 65 patients. Liver Transpl. 2004 Feb;10(2 Suppl 1):S107-10. doi: 10.1002/lt.20036. PMID 14762849
- [Result] Carr BI, Sheetz M, Brown M, et al.: Hepatic arterial 90yttrium-labeled glass microspheres (Therasphere) as treatment for unresectable HCC in forty three patients. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-553, 2002.
- [Result] Carr BI, Brown M, France M, et al.: 90 yttrium labeled glass microspheres in the treatment of hepatocellular carcinoma: initial US experience. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-2346, 2001.